CLINICAL TRIAL: NCT01048918
Title: Characterization of Circulating Tumor Cells (CTC-s) in Patients With Locally Advanced or Metastatic Stage IV Breast Cancer
Status: Completed | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Palo Alto Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08128; CA 111359 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Locally Advanced Breast Cancer; Metastatic (Stage IV) Breast Cancer; Stage III-IV Breast Cancer or Inflammatory
Keywords: Circulating tumor cells in breast cancer
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No Treatment

SUMMARY:
The purpose of this study is to identify tumor cells in the bloodstream (Circulating Tumor Cells, CTC's) from patient's with locally advanced or metastatic (stage IV) breast cancer. Analyzing the tumor is helpful in guiding therapy; however, research has suggested that the number of tumor cells found in the bloodstream (CTC's) signifies more aggressive behavior and increased difficulty in eliminating the cancer. This research will help to develop better ways to treat breast cancer which could be tailored to a patient and may be adjusted to a patient's individual needs.

DETAILED DESCRIPTION:
Up to 60 mL of blood will be collected from each patient at up to 6 time points. Samples will be delivered to the Bruce Laboratory (Palo Alto Research Center) for immunolabeling and FAST scanning. The FAST scanning will utilize CK+, CD45-and DAPI+ labeling as well as cell morphology confirmed by collaborating pathologists to select for CTC with the technology allowing for assessment of up to four additional protein expressions on the surface of CTC's. Additional samples at the proposed time points will be placed on ice and sent over to the Wang Laboratory for the purpose of extracting RNA/microRNA and proteins from CTC's for profiling and further analysis. Benefits are only to society, not the individual. Knowledge obtained from applying the two technologies may help with better selection of therapy, early detection of progression, possibly better diagnosis and development of targeted therapeutic agents in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be > 18 years old.
* Patients are being treated for breast cancer at City of Hope (COH).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Brawerman Center-Outpatient clinics (City of Hope), Pasadena Satellite Office
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2008-09-04 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Targets ER, Her2, and possible M30, VEGFR2, EGFR. Tumor cells found in blood stream. | Blood will be collected at up to 6 time points: Prior to initiating therapy, 8-12 weeks, 20-24 weeks, and at 9,12 and 24 months after initiation of therapy.

SECONDARY OUTCOMES:
Banking leftover blood. Used for future research purposes that have not yet been determined. | Future

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Yuan, MD, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Result] Flores LM, Kindelberger DW, Ligon AH, Cappeletti M, Fiorentino M, Loda M, Cibas ES, Janne PA, Krop IE. Dana-Farber Cancer Institute, Boston, MA; Brigham and Women's Hospital, Boston, MA. Comparison of the Cellsearch Profile Kit (CPK) with the Standard Cellsearch Epithelial Kit (CEK) Demonstrates the CPK Produces Higher Circulating Tumor Cell (CTC) Yields and Is Better Suited for Use in Obtaining CTC's for Molecular Characterization. American Association for Cancer Research 2009; 69(Suppl.): (24). December 15, 2009
- See also: San Antonio Breast Cancer Symposium — http://www.sabcs.org